CLINICAL TRIAL: NCT06347198
Title: A Single-center Exploratory Clinical Study of Oral Inulin in Combination With Fruquintinib Plus Sintilimab as Third- or Further-line Treatment in Metastatic Colorectal Cancer
Brief Title: Oral Inulin in Combination With Fruquintinib Plus Sintilimab as Third- or Further-line Treatment in Metastatic Colorectal Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230807-02
Record Dates: First submitted 2024-03-07; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; inulin; Sintilimab; Fruquintinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; sintilimab; Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Fruquintinib combined with Sintilimab and inulin group) (Experimental)
  Interventions: Drug: Fruquintinib; Drug: Sintilimab; Drug: Inulin
- Control group (Fruquintinib combined with Sintilimab group) (Other)
  Interventions: Drug: Fruquintinib; Drug: Sintilimab

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib: 4 mg/d, qd po, administered continuously for 2 weeks, discontinued for 1 week;
Drug: Sintilimab — Sintilimab: 200 mg, i.v.gtt.D1, administered every 3 weeks;
Drug: Inulin — Inulin: 5g/d, qd po in the first week, 10g/d, bid po from the second week onwards.
  Arms: Intervention group (Fruquintinib combined with Sintilimab and inulin group)

SUMMARY:
This is a single-center exploratory clinical study to explore the efficacy and safety of Oral Inulin in Combination With Fruquintinib Plus Sintilimab as Third- or Further-line Treatment in Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
This was a prospective, two-arm, single-center, exploratory phase I study, randomized 2: 1 into an intervention group (Fruquintinib combined with Sintilimab and inulin group) and a control group (Fruquintinib combined with Sintilimab group). Fruquintinib: 4 mg/d, QD po, administered continuously for 2 weeks with a 1-week discontinuation; Sintilimab 200 mg, I.V., D1, administered every 3 weeks; Inulin: 5 g/d, qd po, in the first week, and 10 g/d, bid po, starting in the second week; Combination therapy was administered every 3 weeks as a treatment cycle. Combination therapy was administered until disease progression, death, or intolerable toxicity.

The study was divided into 3 phases: a screening phase, a treatment phase, and a follow-up phase. Tumor status was assessed using imaging methods every 6 weeks (±7 days) until disease progression (RECIST 1.1) or death (during patient treatment) or intolerable toxicity, and tumor treatment and survival status after disease progression were recorded. Safety observations included changes in AE, laboratory test values, vital signs, and electrocardiographic changes.

ELIGIBILITY:
Inclusion Criteria:

* Have been fully informed about the study and have voluntarily signed an informed consent form;
* Aged 18-75 years (inclusive of 18 and 75 years);
* Pathologically determined unresectable advanced metastatic colorectal cancer;
* Failure of prior second- and back-line standard therapy;
* pMMR or MSS;
* ECOG physical status score of 0-2;
* Expected survival ≥ 6 months;
* Need to have at least one measurable lesion with a maximum diameter of at least 10 mm as determined by spiral CT scanning and at least 20 mm as determined by conventional CT scanning (Criteria for Evaluation of Efficacy in Solid Tumors, i.e., RECIST version 1.1);
* The function of vital organs meets the following requirements (the use of any blood components and cell growth factors is not permitted within *14d prior to enrollment): absolute neutrophil count ≥1.5×10^9/L; platelets ≥75×10^9/L; hemoglobin ≥90g/L; total bilirubin <1.5 times ULN; ALT and/or AST <1.5 times ULN, and for patients with liver metastases <3 times ULN; serum creatinine <1.5 times ULN; endogenous creatinine clearance ≥50 ml/min;
* Men and women of childbearing age need to use effective contraception;
* Not allergic to inulin;
* Subjects agree to provide sufficient blood and fecal samples for immune function and intestinal microbiology testing.

Exclusion Criteria:

* Inability to comply with the study protocol or study procedures;
* Prior treatment with a vascular endothelial growth factor receptor (VEGFR) inhibitor or prior treatment with an immune checkpoint inhibitor;
* Other malignancy within the past 5 years, except for basal or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
* The presence of central nervous system (CNS) metastases or previous brain metastases prior to enrollment
* autoimmune disease or history of autoimmune disease within 4 weeks prior to enrollment
* Previous allogeneic bone marrow transplantation or organ transplantation;
* Uncontrolled malignant ascites (defined as ascites that, in the judgment of the investigator, cannot be controlled by means of diuretics or puncture);
* Severe cardiovascular disease, including unstable angina or myocardial infarction, within 6 months prior to initiation of study treatment, clinically significant cardiovascular disease, including unstable angina or myocardial infarction, within 6 months prior to initiation of study treatment, including, but not limited to, acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months prior to enrollment; congestive Heart failure New York Heart Association (NYHA) classification >2; Ventricular arrhythmia requiring pharmacologic treatment; LVEF (left ventricular ejection fraction) <50%;
* Subjects with hypersensitivity to the study drug or any of its adjuvants;
* Have participated in a clinical trial of another drug not yet approved or marketed in China within 4 weeks prior to enrollment and have been treated with the corresponding trial drug;
* Electrolyte abnormalities of clinical significance as determined by the investigator;
* Pre-existing medically uncontrolled hypertension, defined as systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg;
* The presence of poorly controlled diabetes mellitus (fasting glucose concentration ≥ CTCAE grade 2 after regular treatment) prior to enrollment;
* Any disease or condition that interferes with drug absorption prior to enrollment or the patient is unable to take Fruquintinib orally;
* The presence of gastrointestinal diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresected tumors prior to enrollment, or other conditions that may cause gastrointestinal bleeding or perforation, as determined by the investigator;
* Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding >30 mL within 3 months, vomiting blood, black stool, blood in stool), hemoptysis (>5 mL of fresh blood within 4 weeks), or a thromboembolic event (including stroke events and/or transient ischemic attack) within 12 months;
* Active or uncontrolled serious infection (≥ CTCAE v5.0 grade 2 infection);
* Known human immunodeficiency virus (HIV) infection. Known history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must be excluded from active HBV infection, i.e., HBV DNA-positive (>1×10^4 copies/mL or >2000 IU/ml); known hepatitis C virus infection (HCV) and HCV RNA-positive (>1×10^3 copies/mL)];
* Unresolved toxic reactions above CTCAE v5.0 Grade 1 or higher due to any prior anticancer therapy, excluding alopecia, lymphopenia, and neurotoxicity ≤ Grade 2 due to oxaliplatin;
* Females who are pregnant (positive pregnancy test prior to dosing) or breastfeeding;
* Transfusion therapy, blood products, and hematopoietic factors, such as albumin and granulocyte colony-stimulating factor (G-CSF), received within 14 days prior to enrollment;
* Any other disease with clinically significant metabolic abnormalities, physical examination abnormalities, or laboratory test abnormalities that, in the judgment of the investigator, give reason to suspect that the patient has a disease or condition for which the use of the study medication is inappropriate (e.g., has epileptic seizures that require treatment), or that would interfere with the interpretation of the study results, or that would place the patient at a high level of risk
* Those with routine urinalysis suggestive of urinary protein ≥2+ and a 24-hour urine protein volume >1.0 g;
* Complications requiring long-term immunosuppressive therapy or requiring systemic or topical immunosuppressive corticosteroids (>10 mg/day prednisone or other therapeutic hormones);
* Use of antibiotics or probiotic preparations (probiotic candies, powders, pills, probiotic juices, probiotic yogurts, oligosaccharides, etc.) within the last month
* Patients who, in the opinion of the investigator, are not suitable for enrollment in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Intestinal microbiota diversity, abundance and taxonomic information | 6 months after the recruitment of the last subject.
  Total genomic DNA was extracted from the feces of all patients and metagenomic sequencing was performed. Alpha diversity and beta diversity were used to evaluate the diversity of intestinal microbiota. Abundance and taxonomic information were obtained through taxonomic annotation of the sequencing results.
adverse events | from the date of first dose to the 30 days post the last dose
  Safety will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0.

SECONDARY OUTCOMES:
Objective remission rate (ORR) | 6 months after the recruitment of the last subject.
  was defined as the proportion of patients with the best overall assessment of complete or partial remission. 95% confidence intervals were calculated separately for each group rate using the Clopper-pearson method.
Overall survival (OS) | from date of randomization until the date of progressive disease or EOT due to any cause, assessed up to 1 year
  was defined as the time from enrollment to death from any cause. For patients whose death had not been reported at the time of analysis, the date of their last known survival was used as the censored date.
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  The time (in days) from patient enrollment to disease progression or death.
Disease control rate (DCR) | from date of randomization until the date of progressive disease or EOT due to any cause, assessed up to 1 year
  Disease control rate was defined as the proportion of patients whose best overall assessment was complete remission, partial remission, or stable disease.
Duration of remission (DOR) | from date of the first documentation of response to the date of the first documentation of objective tumor progression or death due to any cause, whichever came first, assessed up to 1 year
  The time interval from the onset of response (when CR or PR is first identified) to progression or death, whichever occurs.
Concentration of various serum metabolites | 6 months after the recruitment of the last subject.
  Use LC-MS/MS to detect and quantify various substances including short-chain fatty acids, bile acids, organic acids, amino acids, sugars, flavonoids, nucleotides, steroid hormones and other substances in serum.
Concentration of various plasma Cytokine Changes | 6 months after the recruitment of the last subject.
  Luminex multi-factor liquid phase analysis technology is used to detect plasma cytokines. The detection indicators include IFN-γ, IL-6, IL-8, IL-10, IL-17A and TNF-α and other cytokines.
Frequency of peripheral blood lymphocyte | 6 months after the recruitment of the last subject.
  Use flow cytometry to detect the frequency of CD4 positive T cells, CD8 positive T cells, natural killer cells, regulatory T cells and other immune cells in peripheral blood.

OTHER OUTCOMES:
Correlation between dietary fiber intake and progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  Patients' dietary fiber intake was collected through dietary questionnaires, and the correlation with progression-free survival was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Min Jin, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No